CLINICAL TRIAL: NCT04444414
Title: Effect of a Manual Therapy Protocol on Balance and Mood States
Brief Title: Manual Therapy on Balance and Mood States
Acronym: MTBMood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID0030
Record Dates: First submitted 2020-06-06; First posted 2020-06-23 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Young Adult
MeSH Terms: interventions — Musculoskeletal Manipulations; Control Groups

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with 2 groups (experimental and control)
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject does not know the group that belonged The evaluator and therapist were different people
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy group (Experimental): Bilateral manipulation lumbosacral, hip joint gapping, stretching the hip rotators with hip and knee flexion, femorotibial gapping, decompression of connective tissue of the patellofemoral region, internal and external joint line opening in laterality, mobilization of the base of the fibula, tibiofibular-talus gapping, and muscle strengthening.
  Interventions: Other: Manual therapy
- Control group (Other): They received no treatment, they just went to the evaluations.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Manual therapy — bilateral manipulation lumbosacral, hip joint gapping, stretching the hip rotators with hip and knee flexion, femorotibial gapping, decompression of connective tissue of the patellofemoral region, internal and external joint line opening in laterality, mobilization of the base of the fibula, tibiofibular-talus gapping, and muscle strengthening.
  Arms: Manual Therapy group
Other: Control group — The control group received no treatment, they only attended the evaluations.
  Arms: Control group

SUMMARY:
The aims of this study was to compare the effectiveness of a protocol of manual therapy on the static balance, dynamic balance and mood states in health participants. This study will consist of a randomized controlled trial. Participants will be healthy subjects divided into 2 groups, being an experimental group that will receive a manual therapy session and a control group without treatment. It will be evaluated at the start of the study, after treatment and one week later.

DETAILED DESCRIPTION:
Background

Evidence suggest that the application of manual therapy could be effective in multiple pathologies, but there are few studies which have investigated the effectiveness of manual therapy in to balance and mood states.

Objective To compare the effectiveness of a protocol of manual therapy on the static balance, dynamic balance and mood states in health participants.

Metods

This is a randomized controlled trial which will be carried out with young adults. The sample will be divided into 2 groups: a) experimental group that will receive a manual therapy session; b) a control group without treatment. All subjects signed the informed consent and confidentiality of the data was reserved according to the Helsinki declaration. The treatments were carried out in the laboratories of the University of Valencia and the project was approved by the institution's ethics committee.

The experimental group to receive manual therapy (Bilateral manipulation lumbosacral, hip joint gapping, stretching the hip rotators with hip and knee flexion, femorotibial gapping, decompression of connective tissue of the patellofemoral region, internal and external joint line opening in laterality, mobilization of the base of the fibula, tibiofibular-talus gapping, and muscle strengthening). The control group will not receive treatment and only evaluations will be performed.

Outcomes

The evaluations will consist of the following variables: Star Excursion Balance Test (SEBT), Unipedal Stance Test (UPST), Patient Global Impression of Change (PGIC) and POMS (Profile Of Mood States). Evaluations will be carried out at three times: at the beginning of the study, after treatment and one week later.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* That they can take all the tests from the study evaluations.

Exclusion Criteria:

* Those who are doing some balance training program.
* Individuals who have some deterioration in balance, regardless of whether the cause is the vestibular system, the visual, proprioceptive, any surgery.
* Participants suffering from tingling or numbness.
* Those who have pain in the lower limbs greater than 3 on the Visual Analog Scale.
* That the lower limbs or in the lumbosacral region have orthopedic problems or traumatic injuries, they will not be able to participate either, including as such scoliosis, ligament pathologies, osteoarthritis, prostheses.
* Pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test (SEBT) | 1-week
  It consists of reaching the lower limb as much as possible, in a standing position, while the other lower limb is kept on a stable support base, at a certain point. The reaches of the leg are evaluated using three determined directions, such as the anterior, the postero-medial and the postero-lateral.

SECONDARY OUTCOMES:
Unipedal Stance Test (UPST) | 1-week
  It consists of a test to measure static balance. Subjects who focus on a fixed point that is marked on the wall and perform the single-legged support. Before lifting the lower limb to be assessed, which will determine the start of the test, the subjects have to cross their arms at chest level, placing their hands on the opposite shoulders. When the subject is ready, close the eyes and raise the lower limb, and the time it is capable of holding is measured with a stopwatch. It is performed later with the other leg
Patient Global Impression of Change (PGIC) | 1-week
  reflects the patient's belief about the effect of the treatment applied. This tool evaluates this perception on a scale that ranges from 1 (the patient is much better) to 7 (the patient is much worse). It also consists of a visual analog scale that classified the improvement from 0 to 10, with the first value being a very good improvement and the second being a significant worsening after treatment.
POMS (Profile Of Mood States) | 1-week
  The POMS is a questionnaire which aims to measure the state of mind. It consists of 58 items, valued using a Likert-type format, with 5 possible response alternatives. From this test, a general index of mood alteration and thirst can be extracted, partially measured: Tension, Depression, Cholera, Vigor, Fatigue and Confusion. Although the POMS has been described as a redundant ladder, it appears to be a multidimensional instrument, with high internal consistency and a relatively stable factor structure.

CONTACTS AND LOCATIONS:
Locations (1):
- Gemma Espí, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Espi-Lopez GV, Serra-Ano P, Vicent-Ferrando J, Sanchez-Moreno-Giner M, Arias-Buria JL, Cleland J, Fernandez-de-Las-Penas C. Effectiveness of Inclusion of Dry Needling in a Multimodal Therapy Program for Patellofemoral Pain: A Randomized Parallel-Group Trial. J Orthop Sports Phys Ther. 2017 Jun;47(6):392-401. doi: 10.2519/jospt.2017.7389. Epub 2017 May 13. PMID 28504067
- [Background] Espi-Lopez GV, Lopez-Martinez S, Ingles M, Serra-Ano P, Aguilar-Rodriguez M. Effect of manual therapy versus proprioceptive neuromuscular facilitation in dynamic balance, mobility and flexibility in field hockey players. A randomized controlled trial. Phys Ther Sport. 2018 Jul;32:173-179. doi: 10.1016/j.ptsp.2018.04.017. Epub 2018 Apr 22. PMID 29793126